CLINICAL TRIAL: NCT03351803
Title: BRCA Founder OutReach (BFOR) Study
Acronym: BFOR
Status: Active, not recruiting | Type: Observational
Sponsor: Memorial Sloan Kettering Cancer Center (Other)
Collaborators: Dana-Farber Cancer Institute (Other); University of Pennsylvania (Other); Beth Israel Deaconess Medical Center (Other); Brigham and Women's Hospital (Other); Breast Cancer Research Foundation (Other); Quest Diagnostics-Nichols Insitute (Industry); LIFELINK.COM INC (Unknown); University of California, Los Angeles (Other)
Responsible Party: Sponsor
Other Study IDs: 17-568
Record Dates: First submitted 2017-11-14; First posted 2017-11-24 (Actual); Last update posted 2025-06-03 (Actual); Status verified 2025-06

CONDITIONS: BRCA1 Mutation; BRCA2 Mutation
Keywords: BRCA; BFOR; Ashkenazi; 17-568

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Participants with Ashkenazi ancestry
  Interventions: Other: BFOR Digital Health solution/Web Portal

INTERVENTIONS:
Other: BFOR Digital Health solution/Web Portal — A digital health solution with Internet-based participant recruitment and ascertainment is a mechanism for distributing access to genetic testing to populations who might not otherwise have access. For this project, LifeLink will build a private web-portal designed by the PI's of the study as described in this protocol, including the wireframes that are in the appendices, that will enable secure contact between study participants and the participating commercial laboratory (Quest Diagnostics) and BFOR researchers, as well as facilitate contacts between study participants and their primary care providers and/or a list of BFOR study centers and BFOR providers.

SUMMARY:
The purpose of this study is to learn how to provide BRCA gene testing to a larger number of people as well as to make testing part of a person's regular medical care.

ELIGIBILITY:
Inclusion Criteria:

* Self-reported age ≥ 25
* Self identify as having at least one of their four grandparents as Ashkenazi Jewish
* Has medical insurance
* Able to understand and read the English-language
* Zip code falls within the catchment areas of the phase of the study (e.g. New York City, Boston, Philadelphia, Los Angeles) accessible to a BFOR designated provider

Exclusion Criteria:

* Under age 25
* No Ashkenazi Jewish ancestry
* Does not have insurance
* Has previously had medical BRCA testing ordered by a health care provider

Min Age: 25 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Participants will be invited to join the BFOR study through information provided to their PCPs by the testing laboratories, and media and community outreach. The study will also be promoted through search engines and by genetics providers who are aware of the study. Approach to the study will be entirely participant-initiated and controlled.
Sampling Method: Non-Probability Sample
Enrollment: 5412 (Actual)
Dates: Start 2017-11-10 (Actual); Primary Completion 2026-05-10 (Estimated); Study Completion 2026-05-10 (Estimated)

PRIMARY OUTCOMES:
Proportion of individuals receiving a standardized program of pretest education who then proceed to genetic testing | Up to 1 year
Proportions of individuals who choose to receive the results through their primary care providers or through the study-provided expert staff | Up to 1 year
Psychosocial impact of genetic population screening utilizing a digital health solution | Up to 1 year
  Quality of life questionnaires measuring cancer-specific distress, perceived risk and BRCA 1/2 testing knowledge will be used.
Facilitators and barriers to engaging primary care providers (PCPs) in the BRCA1/2 results disclosure process | Up to 1 year
  Post-disclosure PCP survey will be used to assess facilitators and barriers in the disclosure process
Participant health updates in personal familial cancer diagnosis and genetic testing depending on method of results communication | Up to 1 year
  Written survey for health and diagnostic updates

CONTACTS AND LOCATIONS:
Overall Officials: Kenneth Offit, MD, MPH, Principal Investigator — Memorial Sloan Kettering Cancer Center
Locations (5):
- United States (5):
  - University of California, Los Angeles, Los Angeles, California
  - Dana Farber Cancer Institute, Boston, Massachusetts
  - Beth Israel Deaconess Medical Center, Boston, Massachusetts
  - Memorial Sloan - Kettering Cancer Center, New York, New York
  - University of Pennsylvania, Philadelphia, Pennsylvania

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Pace LE, Tung N, Lee YS, Hamilton JG, Gabriel C, Revette A, Raja S, Jenkins C, Braswell A, Morgan K, Levin J, Block J, Domchek SM, Nathanson K, Symecko H, Spielman K, Karlan B, Kamara D, Lester J, Offit K, Garber JE, Keating NL. Challenges and Opportunities in Engaging Primary Care Providers in BRCA Testing: Results from the BFOR Study. J Gen Intern Med. 2022 Jun;37(8):1862-1869. doi: 10.1007/s11606-021-06970-8. Epub 2021 Jun 25. PMID 34173196
- [Derived] Pace LE, Lee YS, Tung N, Hamilton JG, Gabriel C, Raja SC, Jenkins C, Braswell A, Domchek SM, Symecko H, Spielman K, Karlan BY, Lester J, Kamara D, Levin J, Morgan K, Offit K, Garber J, Keating NL. Comparison of up-front cash cards and checks as incentives for participation in a clinician survey: a study within a trial. BMC Med Res Methodol. 2020 Aug 17;20(1):210. doi: 10.1186/s12874-020-01086-9. PMID 32807084
- See also: Memorial Sloan Kettering Cancer Center — http://www.mskcc.org